CLINICAL TRIAL: NCT02566642
Title: Patients Preoperative Understanding of the Role of the Anesthesiologist
Brief Title: Understanding the Role of the Anesthesiologist
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: 2013003284
Record Dates: First submitted 2015-09-29; First posted 2015-10-02 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Preoperative Anxiety

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: educational material — pts coming to preadmission testing will view self administered tutorial on the role of anesthesiologist

SUMMARY:
When presenting for elective surgery, patient's often do not completely understand the role that the anesthesiology team plays in their care. In 1999, the American Medical Association (AMA) found that health literacy was a stronger predictor of a person's health than age, income, education level and race. It is very important that the investigators provide information to patients on the role of anesthesiologists in their care before, during, and after the surgery as it has been shown to improve patient anxiety and overall satisfaction.

DETAILED DESCRIPTION:
Background: When presenting for elective surgery, patient's often do not completely understand the role that the anesthesiology team plays in their care. There have been studies done in foreign countries to understand this subject, however, there is a paucity of data in American patients. In 1999, the American Medical Association (AMA) found that health literacy was a stronger predictor of a person's health than age, income, education level and race. It is very important that we provide information to patients on the role of anesthesiologists in their care before, during, and after the surgery as it has been shown to improve patient anxiety and overall satisfaction. The investigators approached 100 patients coming to a pre-admission testing area and asked them to complete an anonymous questionnaire is to understand the extent of patients' knowledge about our roles and to assess where-primary care physician, surgeon, or pre-admission testing clinic-they are being provided this information. Based on the results obtained from this survey we made a targeted effort to improve patient understanding of the role of anesthesiologists. Our goal with this teaching tool is to understand the extent of patients' knowledge about our roles and to assess the efficacy of our pre-admission testing clinic. Based on the results obtained from our prior study we have designed a self administered tutorial on an electronic tablet that will be provided to willing patients during their pre-admission testing clinic visit.

These patients will then be given a short questionnaire on the day of surgery to assess their knowledge and understanding of the care provided to them by the anesthesia team.

Materials and methods: Patients visiting Pre Admission Testing (PAT) in anticipation of surgery will be asked if they wish to volunteer for this study. If so they will be asked to review the 10 question multiple choice tutorial on an electronic tablet. If the patient's response is incorrect the tablet provides the correct response with an explanation. At the PAT visit the patient's name and proposed date of surgery will be obtained. On the day of surgery, these patients will then be given a short questionnaire to assess their knowledge and understanding of the information provided by the tablet exercise. Patients will also be asked to provide demographic information age, gender, race, and highest level of education. Our goal is to obtain 100 anonymous paper surveys. We will compare the survey results of those patients who did not have an opportunity to view the tutorial with those that did to learn whether the tutorial is an effective teaching tool.

Results: All data analysis will be performed using SPSS software (version 16, Chicago, Illinois). Summary statistics, including frequencies and means, will be calculated to describe the sample and to assess the patient population understanding of the role of the anesthesiologists in their care.

Discussion: Based on the results of the first phase of this study, the majority of patients are not fully informed of the role of anesthesiologists. Therefore we have created a self administered tutorial on an electronic tablet which will be administered during their pre-admission testing clinic visit to enhance their understanding of the roles of their anesthesiologist during their surgery.

ELIGIBILITY:
Inclusion Criteria:

* English speaking patients

Exclusion Criteria:

* None

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients coming to the Pre Admission Testing (PAT) at an urban hospital in anticipation of surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Effectiveness of self administered electronic tutorial | day of surgery
  9 point survey comparing the responses from 100 patients who had no intervention to 100 who did

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No